CLINICAL TRIAL: NCT02532842
Title: Paliperidone Palmitate in Early Schizophrenia - A Retrospective, Non-interventional Study of Patients With Newly Diagnosed Schizophrenia Treated With Paliperidone Palmitate Over a 12-Month Period
Brief Title: Non-Interventional Study of Participants With Newly Diagnosed Schizophrenia Treated With Paliperidone Palmitate
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Other Study IDs: CR105892; R092670SCH4041 (Other: Janssen Pharmaceutica NV)
Record Dates: First submitted 2015-08-04; First posted 2015-08-26 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone palmitate
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Schizophrenia: This is a retrospective, non-interventional, multicenter study to retrospectively evaluate hospitalization and medical resource use, patterns of paliperidone palmitate use, and clinical outcomes documented within the medical records of young, adult, newly diagnosed schizophrenia participants for the first 12 months of continuous treatment with paliperidone palmitate. Only retrospective data available from clinical routine practice and documented in a participant's medical record will be collected.

SUMMARY:
The primary objective of this study is to explore hospitalization (number, length and reasons for psychiatric hospitalizations) in young, adult, newly diagnosed schizophrenia participants during the first 12 months of treatment with once monthly paliperidone palmitate in naturalistic clinical settings.

DETAILED DESCRIPTION:
This is a retrospective, non-interventional, multicenter study to retrospectively evaluate hospitalization and medical resource use, patterns of paliperidone palmitate use, and clinical outcomes documented within the medical records of young, adult, newly diagnosed schizophrenia participants for the first 12 months of continuous treatment with paliperidone palmitate. Only retrospective data available from clinical routine practice and documented in a participant's medical record will be collected. The study will be conducted in countries within the EMEA region in which paliperidone palmitate is approved and available. The study will be considered complete with the last data collection for the last participant participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a man or woman aged at least 18 years but not more than 29 years at the time of the first injection of paliperidone palmitate
* Participant must have a documented diagnosis of schizophrenia according to either Tenth Revision of the International Classification of Diseases and Related Health Problems (ICD 10) or Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM 4)
* Participant's first psychotic episode suggestive of schizophrenia must have been clinically evident not longer than 1 year prior to the first injection of paliperidone palmitate
* Participant must have documentation (medical records) of at least 12 months (365 +/- 31 days) continuous treatment with paliperidone palmitate administered for the first time as part of clinical practice. This documentation must have been completed in the participant's records before the initiation of the study site
* Participant must have initiated paliperidone palmitate treatment after the launch date (ie, commercial availability) of paliperidone palmitate at his/her respective site

Exclusion Criteria:

* Participant has either an ICD 10 or DSM 4 axis I diagnosis other than schizophrenia
* Participant was diagnosed with alcohol or drug dependence (except for nicotine and caffeine dependence) according to either ICD 10 or DSM 4 criteria within 1 month prior to initiation of paliperidone palmitate treatment or during the 12 month documentation period
* Participant was treated with any long acting injectable antipsychotic prior to paliperidone palmitate initiation or with a long-acting injectable antipsychotic other than paliperidone palmitate during the 12 month documentation period
* Participant received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 30 days prior to paliperidone palmitate initiation or during the 12 month documentation period
* Participant participated in an interventional or a non-interventional clinical study during the 12 month documentation period

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants with Schizophrenia (according to ICD 10 or DSM IV) who were recently diagnosed (<= 1 year [y] before start of PP treatment) with >= 18 y and <=29 y of age and who received PP for at least 12 months prior to study start of the study (retrospective cohort).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of Hospitalizations | 12 months

SECONDARY OUTCOMES:
Number of Treatment Patterns of paliperidone palmitate as measured by patient records | 12 months
Treatment response Based on clinical illness, symptom severity and measurements of functioning Score | 12 months
Parameters of Psychosocial Functioning based on questionnaire | 12 months
Medical Resource Utilization | 12 months
Psychiatric hospitalizations preceding the first paliperidone palmitate injection | 12 months
Number of Participants with Adverse Events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Janssen Pharmaceutica N.V., Belgium, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (7):
- Croatia (3):
  - Rijeka
  - Split
  - Zagreb
- Russia (2):
  - Moscow
  - Saint Petersburg
- Turkey (Türkiye) (2):
  - Ankara
  - Denizli